CLINICAL TRIAL: NCT05501067
Title: A Tai Chi Training on Hand Grip Strength, Fatigue and Functional Fitness in Post COVID in Elderly Patients.
Brief Title: Tai Chi Training on Hand Grip Strength and Functional Fitness in Post COVID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mohammed Youssef Elhamrawy, Principal Investigator, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Post Covid
Record Dates: First submitted 2022-08-09; First posted 2022-08-15 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Post Covid
MeSH Terms: interventions — Aquatic Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tai chi group (Active Comparator): patients will receive tai chi exercise program
  Interventions: Other: tai chi exercise
- control group (Active Comparator): no intervention
  Interventions: Other: no intervention

INTERVENTIONS:
Other: tai chi exercise — specific tai chi exercise
  Arms: tai chi group
Other: no intervention — no intervention
  Arms: control group

SUMMARY:
to evaluate the effects of participating of Tai Chi program on hand grip strength and Functional Fitness in post Covid

DETAILED DESCRIPTION:
evaluate the effects of Tai Chi and aerobic training on improving hand grip strength, fatigue, and functional fitness in patients with post COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* post covid

Exclusion Criteria:

* medically unstable
* post stroke
* obese
* mentally unstable

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-28 (Estimated)

PRIMARY OUTCOMES:
hand grip strength | 2 months
  dynamometer Handexer HFEH20

SECONDARY OUTCOMES:
functional fitness | 2 months
  senior fitness tests

CONTACTS AND LOCATIONS:
Overall Officials: mohammed elhamrawy, PHD, Principal Investigator — national institute for longevity elderly sciences, Beni Suef University, Egypt
Locations (1):
- National institute for Gerontology, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No